CLINICAL TRIAL: NCT07087834
Title: The Effect of Education Given to Men on Their Perceptions, Attitudes, and Knowledge Levels Toward Cancer Screening
Brief Title: Men's Perceptions, Attitudes, and Knowledge Levels Toward Cancer Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Edanur Özkaya Bozkurt, Research Assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-60116787-020-683945
Record Dates: First submitted 2025-07-04; First posted 2025-07-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Men's Health Screening; Cancer Screening
Keywords: Men's Health; Early Detection of Cancer; Screening
MeSH Terms: interventions — Menogaril

STUDY DESIGN:
Intervention Model Description: After the initial meeting, pre-tests will be administered to the individuals in the experimental group. Subsequently, the days and times of the training sessions will be determined, taking into account the working hours and schedule of the institution and the availability of the employees. The four planned training sessions will then be conducted once a week. The final tests (Cancer Screening Perception Scale, Cancer Screening Attitude Scale, Cancer Screening Knowledge Scale) will be administered to the experimental group one month and three months after the final training session.
  Content and Materials of the Training to be Provided to the Experimental Group The CASEM intervention will be applied to the experimental group. This intervention is an educational intervention consisting of three sessions aimed at increasing men's perceptions, attitudes, and knowledge levels regarding cancer screening. CASEM covers basic information about cancer, common types of cancer among men, screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: CASEM (Cancer Screenings Education for Men)
- Control Group (No Intervention)

INTERVENTIONS:
Other: CASEM (Cancer Screenings Education for Men) — Experimental Group After the initial meeting, pre-tests will be administered to the individuals in the experimental group. Subsequently, the days and times of the training sessions will be determined, taking into account the working hours and schedule of the institution and the availability of the employees. The four planned training sessions will then be conducted once a week. The post-test (Cancer Screening Perception Scale, Cancer Screening Attitude Scale, Cancer Screening Knowledge Scale) will be administered to the experimental group one month and three months after the final training session.
  Content and Materials of the Training to Be Provided to the Experimental Group The intervention described in the appendix will be applied to the experimental group. This intervention is an educational intervention consisting of three sessions aimed at increasing men's perceptions, attitudes, and knowledge levels regarding cancer screening. ... It covers basic information about cancer, commo
  Arms: Experimental group

SUMMARY:
Countries are establishing national and international cancer control programs in response to cancer, which has become a global problem. Therefore, cancer is a disease that can be combated not only through investments in treatment, but also through efforts focused on prevention and early diagnosis. According to GLOBOCAN 2022 data, more than 51% of all cancer cases worldwide occur in men. The three most common types of cancer in men are lung cancer, prostate cancer, and colorectal cancer. Increasing awareness, attitudes, and knowledge levels regarding cancer screenings, especially for preventable diseases, will increase participation in screening programs. Increased knowledge levels will translate into positive health behaviors. This study will be conducted as a randomized controlled trial to determine the effect of the Cancer Screenings Education for Men (CASEM) intervention on men's perceptions, attitudes, and knowledge regarding cancer screening programs. Research data will be collected at a public institution between September 2025 and September 2026. The study sample will consist of a total of 78 male individuals, including 39 experimental and 39 control groups that meet the inclusion criteria. Male individuals will be assigned to the experimental and control groups using stratified randomization. The Individual Identification Form, Cancer Screening Perception Scale, Cancer Screening Attitude Scale, and Cancer Screening Knowledge Scale will be used. IBM SPSS 29.0 software will be used to analyze the data obtained from the study. This study will be an important one that addresses Turkey's future vision within the scope of the Twelfth Development Plans and supports the goals and policy measures of the development plan. In addition, our study serves the Sustainable Development Goals, which are among the most important global goals in the context of sustainability. It is expected to have implications for health practices and planning.

ELIGIBILITY:
In Turkey, the National Cancer Screening Program for men involves a fecal occult blood test every two years for those aged 50-70 and a colonoscopy every 10 years. Although men under the age of 50 are not included in the routine screening program, there are many simple screening methods for various cancers. After reviewing the literature and considering the current prevalence of cancer, it was decided that men aged 30 and older are suitable for sampling. The inclusion criteria for the study were determined in accordance with the relevant literature (Abasi et al., 2021; Echeverri et al., 2022; Makarov et al., 2021; Vernon et al., 2024).

Inclusion criteria

To be included in the study, participants must meet all of the following criteria:

* Be 30 years of age or older at the time of the study,
* Be at least literate,
* Have no cognitive, visual, or orthopedic impairments that would prevent them from completing the questionnaires,
* Be able to speak and understand Turkish,
* Have no previous history of cancer diagnosis or cancer treatment,
* Agree to participate in the study.

Exclusion criteria

Participants are excluded from the study if they meet any of the following criteria:

* Having previously had cancer and undergone cancer treatment,
* Not currently employed at the institution (e.g., on temporary assignment),
* Refusing to participate in the study.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The change in the cancer screening perception of the experimental group according to the Cancer Screening Perception Scale scores at the end of the first and third month | 3 months
  It is a 26-item scale developed by Mahmood et al. (2016). Its validity and reliability in Turkish were established by Bozkurt and Yılmaz (2024). The scale items generally cover. The scale has five sub-factors: "Perceived Severity, Perceived Sensitivity, Perceived Benefits, Perceived Barriers, and Action Cues." The scale is a 6-point Likert scale (1 = Strongly disagree, 6 = Strongly agree). To prevent confusion, there is no "undecided" option. The scale is not aggregatable, and each sub-dimension in the scale is evaluated separately.
The change in the cancer screening attitude of the experimental group according to the Cancer Screening Attitude Scale scores at the end of the first and third month | 3 months
  The scale was developed by Yıldırım-Öztürk and colleagues (2020). The scale consists of 24 items and a single dimension. The scale is a five-point Likert scale. The items comprising the scale are answered on a scale ranging from 5 to 1, as follows: "5: I completely agree, 4: I somewhat agree, 3: I neither agree nor disagree, 2: I somewhat disagree, 1: I completely disagree." The scale is suitable for use on women and men aged 30-70 who are at least literate and do not have cognitive, visual, or orthopedic impairments that would prevent them from completing the scale.
The change in the cancer screening knowledge of the experimental group according to the Cancer Screening Knowledge Scale scores at the end of the first and third month | 3 months
  The scale was developed by Yıldırım-Öztürk and Uyar (2023). The scale consists of 25 items and 3 subscales. The subscales of the scale have not been specifically named. The first subscale of the scale consists of 10 items (items 8, 17-23, 25, and 28), the second subscale consists of 9 items (items 4, 5, 7, 10, 12, 13, 15, 16, and 27), and the third subscale has 6 items (items 1-3, 9, 11, 24). The scale is a three-point rating scale. The scale is answered on a scale from 1 to 3, with "1: Correct, 2: Incorrect, 3: I don't know." When calculating the scale score, "True" responses are scored as 1 point, while 'False' and "I don't know" responses are scored as 0 points. The lowest possible score on the scale is 0, and the highest possible score is 25. When calculating the scale score, the three items with negative meanings (Items 2, 11, and 24) must be reverse-coded. No cutoff point has been established for the scale score.

SECONDARY OUTCOMES:
Individuals' status regarding cancer screening in the final test conducted at the end of the third month after education | 3 months
  Both groups will be asked whether they conducted cancer screening in their final tests. A single-question survey will be administered, asking, "Have you had a cancer screening in the last three months?" Responses will be evaluated on a two-point Likert scale, with options for 'yes' and "no."

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will share.
Supporting Information: Study Protocol, SAP
Time Frame: starting 1 months after publication
Access Criteria: all people access